CLINICAL TRIAL: NCT02436473
Title: Clinical Efficacy of Fluoride Toothpastes Using an In Situ Caries Model
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was cancelled. No subjects were enrolled and no data has been collected
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 203161
Record Dates: First submitted 2015-05-04; First posted 2015-05-06 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test fluoride toothpaste (Experimental): Participants will apply 1.5 weighed g (± 0.1 g) of the study toothpaste to a wet toothbrush and brush their natural teeth twice daily for one timed minute. Participants will wear their mandibular partial denture with test specimens while brushing and continuously for 24 hours a day during each of the 4-week treatment periods
  Interventions: Drug: Toothpaste containing 1150ppm F
- Fluoride free (0ppm F) reference control toothpaste (Placebo Comparator): Participants will apply 1.5 weighed g (± 0.1 g) of the study toothpaste to a wet toothbrush and brush their natural teeth twice daily for one timed minute. Participants will wear their mandibular partial denture with test specimens while brushing and continuously for 24 hours a day during each of the 4-week treatment periods.
  Interventions: Other: Toothpaste containing 0ppm F
- Low dose fluoride (250ppm F) reference control toothpaste (Active Comparator): Participants will apply 1.5 weighed g (± 0.1 g) of the study toothpaste to a wet toothbrush and brush their natural teeth twice daily for one timed minute. Participants will wear their mandibular partial denture with test specimens while brushing and continuously for 24 hours a day during each of the 4-week treatment periods.
  Interventions: Drug: Toothpaste containing 250ppm F
- Fluoride (1150ppm F) reference control toothpaste (Active Comparator): Participants will apply 1.5 weighed g (± 0.1 g) of the study toothpaste to a wet toothbrush and brush their natural teeth twice daily for one timed minute. Participants will wear their mandibular partial denture with test specimens while brushing and continuously for 24 hours a day during each of the 4-week treatment periods.
  Interventions: Drug: Toothpaste containing 1150ppm F

INTERVENTIONS:
Drug: Toothpaste containing 1150ppm F — US marketed toothpaste containing 1150ppm of F
  Arms: Test fluoride toothpaste
Other: Toothpaste containing 0ppm F — Experimental toothpaste containing 0ppm F
  Arms: Fluoride free (0ppm F) reference control toothpaste
Drug: Toothpaste containing 250ppm F — Experimental toothpaste containing 250ppm F
  Arms: Low dose fluoride (250ppm F) reference control toothpaste
Drug: Toothpaste containing 1150ppm F — Experimental toothpaste containing 1150ppm F
  Arms: Fluoride (1150ppm F) reference control toothpaste

SUMMARY:
The purpose of this study is to evaluate the effect of the test toothpaste containing 1150 parts per million (ppm) of fluoride (F) on the mineral content of demineralized enamel specimens, in an in situ caries model system, by comparing the differences in net remineralization change (ΔM) following use of the test toothpaste with a fluoride free (0 ppm F) reference control toothpaste.

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrates understanding of the study.
2. Aged 18 to 85 years.
3. Understands and is willing, able and likely to comply with all study procedures and restrictions.
4. Has good general health (in the opinion of the investigator or medically qualified designee).
5. Currently living in the Indianapolis, Indiana area.
6. Currently wearing a removable mandibular partial denture with sufficient room in the posterior buccal flange area to accommodate two enamel specimens.
7. Have no current active caries or periodontal disease and all restorations in a good state of repair.
8. Have a salivary flow rate in the range of normal values.

Exclusion Criteria:

1. Pregnant or breast feeding women.
2. Known or suspected intolerance or hypersensitivity to the study materials or their stated ingredients.
3. Currently taking antibiotics or have taken antibiotics in the two weeks prior to the screening visit.
4. Unable to measure product weights accurately using the assigned study scale as determined by the study staff as demonstrated.
5. Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
6. Have received a professional fluoride treatment within 14 days of randomization to the first treatment.
7. Recent history (within the last year) of alcohol or other substance abuse.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Net remineralization change (ΔM) of demineralised enamel specimens following use of the test toothpaste with a fluoride free reference control toothpaste | 4 weeks
  The change in mineral content (ΔM) of the lesions as measured by Transverse Microradiography (TMR) will be calculated by the following formula: ΔM= (Post-treatment ΔZ - baseline ΔZ)

SECONDARY OUTCOMES:
Net remineralization change (ΔM) of demineralised enamel specimens following use of the test toothpaste with all other treatments | 4 weeks
  The change in mineral content (ΔM) of the lesions as measured by TMR will be calculated by the following formula: ΔM= (Post-treatment ΔZ - baseline ΔZ)
Changes in enamel lesion depth (ΔL) following use of the test toothpaste with all other treatments | 4 weeks
  The change in lesion depth (ΔL) as measured by TMR will be calculated by: ΔL= (Post-treatment lesion depth - baseline lesion depth)
Net change in surface zone mineral content (ΔSZmax) following use of the toothpaste with all other treatments | 4 weeks
  The change in SZmax (ΔSZmax) as measured by TMR will be calculated by: ΔSZmax= (Post-treatment SZmax - baseline SZmax)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline